CLINICAL TRIAL: NCT00439023
Title: Effect of Glucose in Dialysis Water on Blood Pressure and Vasoactive Hormones in Dialysis Patients
Brief Title: Glucose in Dialysis Water in Non-diabetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MED.RES.2007.01.EBP
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2007-09

CONDITIONS: Renal Failure, Chronic
Keywords: Chronic renal failure, dialysis, hemodialysis,
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dialysis; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: dialysis with glucose in dialysis water

SUMMARY:
The purposes are

1. to measure the effect of dialysis with glucose on blood pressure, pulse rate, plasma concentration of glucose, plasma concentrations of glucagon, growth hormone, renin, angiotensin II, endothelin and body temperature, and
2. to analysis the relationship between changes in blood pressure on the one hand and changes in vasoactive hormones on the other

DETAILED DESCRIPTION:
Measurement of hormones and blood pressure during dialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years,
2. Both men and women,
3. Dialysis treatment for at least three months

Exclusion Criteria:

1. Heart failure,
2. Chronic liver disease,
3. Diabetes mellitus,
4. Malignant disease,
5. Nephrotic syndrome,
6. Lack of compliance, 7 Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Effect of glucose in dialysis water on blood pressure, insulin and vasoactive hormones | one week

SECONDARY OUTCOMES:
Relationship between changes in blood pressure and changes in hormones during treatment | one week

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Regional Hospital Holstebro
Locations (1):
- Holstebro Hospital, Holstebro, Denmark